CLINICAL TRIAL: NCT06781892
Title: Strategies for Defibrillation During Out-of-Hospital Cardiac Arrest - A Randomized Clinical Trial
Brief Title: Strategies for Defibrillation During Out-of-Hospital Cardiac Arrest
Acronym: STRAT-DEFI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lars Wiuff Andersen (Other)
Collaborators: University of Aarhus (Other)
Responsible Party: Sponsor-Investigator, Lars Wiuff Andersen, Professor, Aarhus University Hospital
Organization: Aarhus University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 00006
Record Dates: First submitted 2025-01-14; First posted 2025-01-17 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Cardiac Arrest (CA)
Keywords: Out-of-hospital cardiac arrest; Defibrillation; Double-sequential defibrillation
MeSH Terms: conditions — Heart Arrest; Out-of-Hospital Cardiac Arrest

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Anterior-lateral pad positioning (Active Comparator)
  Interventions: Other: Anterior-lateral pad positioning
- Anterior-posterior pad positioning (Experimental)
  Interventions: Other: Anterior-posterior pad positioning
- Double-sequential defibrillation (Experimental): Anterior-lateral pad positioning combined with anterior-posterior pad positioning for a total of 4 pads and 2 shocks.
  Interventions: Other: Double-sequential defibrillation

INTERVENTIONS:
Other: Anterior-lateral pad positioning — Defibrillation pads positioned anterior-lateral
  Arms: Anterior-lateral pad positioning
Other: Anterior-posterior pad positioning — Defibrillation pads positioned anterior-posterior
  Arms: Anterior-posterior pad positioning
Other: Double-sequential defibrillation — Combination of anterior-lateral and anterior-posterior pad positioning for a total of 4 pads and 2 shocks.
  Arms: Double-sequential defibrillation

SUMMARY:
The "Strategies for Defibrillation during Out-of-Hospital Cardiac Arrest" (STRAT-DEFI) trial is an investigator-initiated, individually randomized, 3-group clinical trial comparing standard anterior-lateral pad positioning with anterior-posterior positioning and double sequential defibrillation during adult out-of-hospital cardiac arrest.

ELIGIBILITY:
Inclusion Criteria:

1. Out-of-hospital cardiac arrest
2. Age ≥ 18 years
3. ≥ 1 manual defibrillation attempt by emergency medical services
4. Shockable rhythm as the last known rhythm
5. Two manual defibrillators present on-site

Exclusion Criteria:

1. Blunt trauma, penetrating trauma, or burn injury suspected to be the cause of the cardiac arrest
2. Prior enrollment in the trial
3. Posterior pad placement not deemed possible by on-site clinician

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 909 (Estimated)
Dates: Start 2025-03-15 (Actual); Primary Completion 2028-03-01 (Estimated); Study Completion 2029-03-01 (Estimated)

PRIMARY OUTCOMES:
Survival at 30 days | 30 days after the cardiac arrest

SECONDARY OUTCOMES:
Survival at 90 days | 90 days after the cardiac arrest
Favorable neurological outcome at 30 days | 30 days after the cardiac arrest
  Neurological outcome will be assessed with the modified Rankin Scale (mRS) which is a scale from 0 to 6 assessing neurological/functional outcomes after brain damage with higher scores indicating worse neurological/functional outcomes. The scale will will be dichotomized as favorable (mRS 0-3) vs. unfavorable (mRS 4-6).
Favorable neurological outcome at 90 days | 90 days after the cardiac arrest
  Neurological outcome will be assessed with the modified Rankin Scale (mRS) which is a scale from 0 to 6 assessing neurological/functional outcomes after brain damage with higher scores indicating worse neurological/functional outcomes. The scale will will be dichotomized as favorable (mRS 0-3) vs. unfavorable (mRS 4-6).

CONTACTS AND LOCATIONS:
Locations (6):
- Denmark (6):
  - Emergency Medical Services, the North Denmark Region, Aalborg
  - Danish Air Ambulance, Danish Regions, Aarhus N
  - Prehospital Emergency Medical Services, Central Denmark Region, Aarhus N
  - Copenhagen Emergency Medical Services, the Capital Region of Denmark, Ballerup Municipality
  - The Prehospital Center, Region Zealand, Næstved
  - Emergency Medical Services, the Region of Southern Denmark, Vejle

IPD SHARING:
Plan to Share IPD: Yes
De-identified data. All relevant trial-related documents, including the protocol, data dictionary, and the main statistical code, will be shared along with the data.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: After publication of the last results (i.e., 1-year follow-up), all de-identified individual patient data will be made available for data sharing as allowed within Danish law. There will be no predetermined end date for the data sharing.
Access Criteria: Data will be available for any research purpose to all interested parties who have approval from an independent review committee if required and who have a methodological sound proposal as determined by the steering committee of the current trial. Only the methodological qualities and not the purpose or objective of the proposal will be considered. Interested parties will be able to request the data by contacting the principal investigator.